CLINICAL TRIAL: NCT03782922
Title: Effect of an Exercise Training Programm on Mental and Anatomical Characteristics of Physiotherapy Students - a Randomized Controlled Trial
Brief Title: Exercise Training Programm for Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: THIM - die internationale Hochschule für Physiotherapie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018-01954
Record Dates: First submitted 2018-12-05; First posted 2018-12-20 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2018-12

CONDITIONS: Healthy; Student; Physical Therapy
Keywords: exercise; anatomical; mental; training program
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Program (Experimental)
  Interventions: Other: Exercise Training Program
- Control (No Intervention)

INTERVENTIONS:
Other: Exercise Training Program — 10min of coordination and strength training (2-3x per week) during 2-6 weeks
  Arms: Exercise Training Program

SUMMARY:
In this study, i.e. randomized controlled trial, the effect of an exercise training program on mental and anatomical characteristics of physiotherapy students is measured.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18
* signed consent
* THIM student
* good health status

Exclusion Criteria:

* alcohol
* drugs
* smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
d2-R-Test | Change from baseline attention and concentration at 4 weeks (objective)
  Mental
AKA-Questionnaire (attention, concentration, learning ability) | Change from baseline attention and concentration at 4 weeks (subjective)
  Participants fill out a questionnaire about attention, concentration and learning ability. There are five possible answers for each item from 1 (completely disagree) to 5 (completely agree).
M360 - physiological parameter of the spine | Change from baseline position and mobility of the spine at 4 weeks
  Participants are measured in different positions (upright, flexion, extension; measured in degrees) to assess position, stability and mobility of the spine. The M360 will be guided along the back and the data will be collected electronically (https://www.idiag.ch/idiag-m360/).
Pain (Visual Analogue Scale) | Change from baseline pain (back) at 4 weeks
  Participants can use this scale to classify their pain from "No pain" and "Maximum pain imaginable" by means of a slider.
FAW-Questionnaire (Actual physical well-being) | Change from baseline physical well-being at 4 weeks
  Participants fill out a questionnaire with 58 questions. Each question has five possible answers from 0 (completely disagree) to 4 (completely agree). The highter the score the better the actual physical well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- THIM University of Applied Sciences, Landquart, Switzerland